CLINICAL TRIAL: NCT07032558
Title: A Randomized, Open-label, Single Oral Dose, Two-period, Cross-over Trial to Evaluate the Pharmacokinetics of Pelubiprofen-Tramadol (DW-1021) Controlled Release Film Coated Tablets (Pelubiprofen 45mg-Tramadol 45.9mg Salt) (Test Drug) in Comparison With the Co-administration of Each of Pelubi CR 45mg Controlled Release Film Coated Tablets (Pelubiprofen 45mg) and Zytram CR 75mg Controlled Release Film Coated Tablets (Tramadol HCl 75mg) in Healthy Adult Vietnamese Male Subjects Under Fasting Condition
Brief Title: Comparison of DW-1021 and Separate Doses of Pelubi CR and Zytram CR Under Fasting Conditions
Acronym: DW-1021
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Haiphong University of Medicine and Pharmacy (Other)
Collaborators: Daewon Pharmaceutical Co., Ltd. (Industry); Big Leap Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW-1021; Protocol No. DW-1021 (Other: Daewon Pharmaceutical Co., Ltd.)
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteer
Keywords: Pelubiprofen; Tramadol; DW-1021; Pharmacokinetics; Fixed-Dose Combination; Bioavailability
MeSH Terms: interventions — pelubiprofen; Tramadol

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label, single-dose, 2-treatment, 2-period, 2-sequence (2x2) crossover study conducted under fasting conditions. Fourteen healthy male volunteers will be randomly assigned to one of two sequences: Test-Reference (Group A) or Reference-Test (Group B), with a 14-day washout period between dosing periods. The test drug (DW-1021, Pelubiprofen 45 mg - Tramadol 45.9 mg salt) or the reference drugs (Pelubi CR 45 mg and Zytram CR 75 mg) will be administered orally with 150 mL of water after at least 10 hours of fasting. Blood samples will be collected up to 48 hours post-dose in each period for pharmacokinetic evaluation.
Masking Description: This is an open-label study. No parties are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A: Test → Reference (Experimental): Participants in this arm will receive the test drug DW-1021 (Pelubiprofen 45 mg - Tramadol 45.9 mg salt) in Period I, followed by the reference drugs-Pelubi CR 45 mg and Zytram CR 75 mg-in Period II. A 14-day washout period separates the two dosing periods.
  Interventions: Drug: DW-1021; Drug: Pelubi CR + Zytram CR
- Sequence B: Reference → Test (Active Comparator): Participants in this arm will receive the reference drugs-Pelubi CR 45 mg and Zytram CR 75 mg-in Period I, followed by the test drug DW-1021 (Pelubiprofen 45 mg - Tramadol 45.9 mg salt) in Period II. A 14-day washout period separates the two dosing periods.
  Interventions: Drug: DW-1021; Drug: Pelubi CR + Zytram CR

INTERVENTIONS:
Drug: DW-1021 — DW-1021 is a fixed-dose combination tablet containing Pelubiprofen 45 mg and Tramadol 45.9 mg (as a salt), formulated as a controlled-release film-coated tablet. It is administered as a single oral dose with 150 mL of water under fasting conditions for the evaluation of pharmacokinetics in healthy adult male volunteers.
  Other Names: Pelubiprofen 45 mg - Tramadol 45.9 mg salt combination; Pelubiprofen-Tramadol fixed-dose combination
Drug: Pelubi CR + Zytram CR — The reference treatment consists of two separate controlled-release film-coated tablets: Pelubi CR (Pelubiprofen 45 mg) and Zytram CR (Tramadol HCl 75 mg). These are co-administered as a single oral dose with 150 mL of water under fasting conditions to compare the pharmacokinetic profile against the fixed-dose combination DW-1021.
  Other Names: Pelubiprofen 45 mg controlled-release tablet; Tramadol HCl 75 mg controlled-release tablet

SUMMARY:
This is a Phase 1, randomized, open-label, single-dose, two-period, cross-over study to evaluate the pharmacokinetics (PK) of DW-1021, a fixed-dose combination tablet containing Pelubiprofen 45 mg and Tramadol 45.9 mg (as a salt), in healthy adult Vietnamese male volunteers. The study compares DW-1021 with the co-administration of two reference drugs: Pelubi CR 45 mg (Pelubiprofen) and Zytram CR 75 mg (Tramadol HCl), under fasting conditions.

A total of 14 eligible participants will be randomly assigned to receive either the test drug followed by the reference drugs, or vice versa, with a 14-day washout period between the two dosing periods. Blood samples will be collected over a 48-hour period after each administration to evaluate drug concentrations. The main purpose is to assess and compare the rate and extent of absorption (Cmax, AUC) of the test and reference products.

The study is sponsored by Haiphong University of Medicine and Pharmacy in collaboration with Daewon Pharmaceutical Co., Ltd. It is conducted under ethical approval by the National Ethics Committee in Biomedical Research of Vietnam.

DETAILED DESCRIPTION:
This clinical trial is designed to evaluate and compare the pharmacokinetic characteristics of DW-1021, a fixed-dose combination of Pelubiprofen and Tramadol in salt form (Pelubiprofen 45 mg - Tramadol 45.9 mg), with the co-administration of the individual components-Pelubi CR 45 mg (controlled release Pelubiprofen) and Zytram CR 75 mg (controlled release Tramadol hydrochloride)-in healthy adult male Vietnamese volunteers under fasting conditions.

This is an open-label, randomized, single-dose, two-treatment, two-period, two-sequence crossover study. Fourteen eligible participants will be randomized into two sequences: Test-Reference (TR) and Reference-Test (RT), with each dosing period separated by a 14-day washout. Study drugs will be administered in a fasted state, and blood samples will be collected at multiple time points up to 48 hours post-dose for pharmacokinetic analysis.

The primary PK parameters include Cmax and AUCt. Secondary PK parameters include Tmax, AUC∞, and t1/2. Safety will be monitored through assessment of adverse events, vital signs, clinical laboratory tests, and physical examinations throughout the study.

The trial is sponsored by Haiphong University of Medicine and Pharmacy. Analytical testing of plasma concentrations will be performed by Invites Bio-Core, and CRO support is provided by Big Leap Clinical Research Support JSC. The study is approved by the National Ethics Committee in Biomedical Research of Vietnam (Approval No. 277/CN-HĐĐĐ, dated 12/12/2024). This study was additionally approved for protocol amendments by the Vietnamese Ministry of Health under Decision No. 3840/QĐ-BYT, dated December 19, 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged 20 to 40 years at screening visit
2. Body Mass Index (BMI) between 18.5 and 24.9 kg/m²
3. Body weight greater than 50 kg
4. Systolic blood pressure between 100 mmHg and 129 mmHg; diastolic blood pressure less than 84 mmHg
5. Regular heart rate ranging from 60 to 90 beats per minute
6. No clinically significant medical history or evidence of congenital or chronic diseases, including but not limited to: hypertension, orthostatic hypotension, hypoglycemia when fasting, swallowing difficulties, diabetes, cardiovascular diseases, pulmonary diseases, gastrointestinal diseases, liver insufficiency, renal insufficiency, endocrine disorders, neurological or psychiatric disorders, immunological, hematological, or hereditary diseases, tuberculosis, or infectious diseases
7. Suitable laboratory test results (hematology, urinalysis, blood chemistry, HCV/AIDS, HBsAg, anti-HCV) and electrocardiogram (ECG) at screening: no pathological findings; clinical laboratory parameters within the normal range or, if outside the normal range, not clinically significant as judged by the investigator
8. Willing and able to provide written informed consent after being fully informed about the study objectives and possible adverse effects
9. Agree to use effective contraception from initial administration until 7 days after the last dose of test or reference drugs

Exclusion Criteria:

1. Use of drugs that induce or inhibit drug-metabolizing enzymes (e.g., barbiturates) within 30 days prior to administration, or use of any medication that might affect the study within 10 days prior to administration
2. Participation in any other clinical trial within 3 months prior to screening
3. Blood donation within 8 weeks prior to drug administration
4. History of gastrointestinal surgery that may affect drug absorption
5. History of drug abuse, or use of alcohol, drugs, or tobacco products within 1 year before participation
6. Known hypersensitivity or allergy to the test or reference drug or their components
7. Known genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption, which are characterized by symptoms like diarrhea and bloating after consuming dairy products
8. Suffering from dysphagia

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 0 to 48 hours post-dose in each period
  Cmax represents the peak plasma concentration of the drug after administration. It is used to compare the rate of absorption between the test and reference products.
Area under the plasma concentration-time curve from time 0 to the last measurable concentration (AUCt) | 0 to 48 hours post-dose in each period
  AUCt is a pharmacokinetic parameter representing the total drug exposure from administration to the last quantifiable time point. It is used to compare the extent of absorption between DW-1021 and the reference drugs.

SECONDARY OUTCOMES:
Area under the curve extrapolated to infinity (AUC∞) | 0 to 48 hours post-dose in each period
  AUC∞ represents the total drug exposure over time, extrapolated beyond the last measured concentration. It helps assess complete systemic exposure.
Terminal elimination half-life (t1/2) | 0 to 48 hours post-dose in each period
  The time it takes for the plasma concentration of the drug to decrease by 50%. It is used to understand the drug elimination kinetics.
Time to reach maximum plasma concentration (Tmax) | 0 to 48 hours post-dose in each period
  Tmax is defined as the time point at which the maximum plasma drug concentration is observed following drug administration. It is used to compare the absorption rate between DW-1021 and the reference products.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial and Bioequivalence Center, Haiphong, Hai Phong, Vietnam

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and the limited scope of the Phase I pharmacokinetic study in healthy volunteers. The study does not include plans or infrastructure for external data sharing.

REFERENCES:
- [Background] Choi IA, Baek HJ, Cho CS, Lee YA, Chung WT, Park YE, Lee YJ, Park YB, Lee J, Lee SS, Yoo WH, Song JS, Kang SW, Kim HA, Song YW. Comparison of the efficacy and safety profiles of a pelubiprofen versus celecoxib in patients with rheumatoid arthritis: a 6-week, multicenter, randomized, double-blind, phase III, non-inferiority clinical trial. BMC Musculoskelet Disord. 2014 Nov 18;15:375. doi: 10.1186/1471-2474-15-375. PMID 25403311
- [Background] Shin JS, Baek SR, Sohn SI, Cho YW, Lee KT. Anti-inflammatory effect of pelubiprofen, 2-[4-(oxocyclohexylidenemethyl)-phenyl]propionic acid, mediated by dual suppression of COX activity and LPS-induced inflammatory gene expression via NF-kappaB inactivation. J Cell Biochem. 2011 Dec;112(12):3594-603. doi: 10.1002/jcb.23290. PMID 21809372